CLINICAL TRIAL: NCT06870435
Title: Comparison and Strategy Optimization of Plasma Epstein-Barr Virus (EBV) DNA and BNLF2b Total Antibodies (P85-Ab) with VCA-IgA and EBNA1-IgA for Screening Nasopharyngeal Carcinoma in High-risk Areas
Brief Title: Comparison and Strategy Optimization of Plasma EBV DNA and P85-Ab with VCA/EBNA1-IgA for Screening Nasopharyngeal Carcinoma in High-risk Areas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ming-Yuan Chen (Other)
Responsible Party: Sponsor-Investigator, Ming-Yuan Chen, Professior, Chief physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ZDWY.BYAFZZX.032
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-01

CONDITIONS: Nasopharyngeal Carcinoma (NPC); Screening; Epstein Barr Virus
Keywords: Nasopharyngeal Carcinoma (NPC); Screening; Epstein Barr Virus; EBV DNA; EBV antibody
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Epstein-Barr Virus Infections | interventions — Blood Specimen Collection; Biopsy

STUDY DESIGN:
Intervention Model Description: All participants will be tested for Epstein-Barr virus (EBV) associated biomarkers, including the two-antibody method (VCA-IgA and EBNA1-IgA), BNLF2b total antibodies (P85-Ab), and plasma EBV DNA. Furthermore, novel screening biomarkers, such as next-generation sequencing for EBV and castoff cells using nasopharyngeal swabs, will be explored.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Screening cohort (Experimental): Participants aged between 30 and 69 years old.
  Interventions: Biological: Blood, nasopharyngeal swab and saliva; Diagnostic Test: EBNA1-IgA, VCA-IgA, P85-Ab and EBV DNA; Diagnostic Test: Novel screening biomarkers; Diagnostic Test: Endoscopic examinations with or without biopsy

INTERVENTIONS:
Biological: Blood, nasopharyngeal swab and saliva — Collect blood, nasopharyngeal swab and saliva samples from participants.
Diagnostic Test: EBNA1-IgA, VCA-IgA, P85-Ab and EBV DNA — Detect EBNA1-IgA, VCA-IgA, P85-Ab and EBV DNA for all participants.
Diagnostic Test: Novel screening biomarkers — Next-generation sequencing for EBV and castoff cells using nasopharyngeal swabs, etc..
Diagnostic Test: Endoscopic examinations with or without biopsy — High-risk participants will refer to endoscopic examinations with or without biopsy

SUMMARY:
This study is a prospective, self-controlled, multicenter clinical trial. All participants will be tested for Epstein-Barr virus (EBV) associated biomarkers, including the two-antibody method (VCA-IgA and EBNA1-IgA), BNLF2b total antibodies (P85-Ab), and plasma EBV DNA. Furthermore, novel screening biomarkers, such as next-generation sequencing for EBV and castoff cells using nasopharyngeal swabs, will be explored.

First, it aims to investigate whether plasma EBV DNA testing or the P85-Ab testing can achieve higher sensitivity than the current standard two-antibody method testing while maintaining specificity in NPC screening, thereby identifying the optimal initial NPC screening strategy. Based on the determined optimal initial screening strategy, the study will validate the proposed two-step method (subjects first undergo two-antibody method testing and P85-Ab testing; those positive for either one biomarker above proceed to plasma EBV DNA testing; subjects positive in both steps are defined as high-risk and receive endoscopic examinations with or without biopsy) compared with the single-step method (subjects simultaneously undergo two-antibody method testing, P85-Ab testing, and plasma EBV DNA testing; subjects with any positive biomarker undergo endoscopic examinations with or without biopsy) and each single screening testing. The aim is to determine whether two-step method can further improve the positive predictive value (PPV) while maintaining non-inferior sensitivity, thereby enhancing screening efficiency, reducing the rate of invasive procedures (such as endoscopic biopsies), and lowering medical costs and insurance burdens.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent.
* Age between 30 and 69 years at the time of screening.
* Residents of Guangdong Province or Guangxi Province.
* Able to cooperate with long-term follow-up.

Exclusion Criteria:

* Severe medical comorbidities, significant organ (heart, lung, liver, kidney) dysfunction, or psychiatric disorders.
* Severe autoimmune diseases or immunodeficiency.
* History of or current malignant tumors.
* Inability to cooperate with the study due to psychological, social, familial, or geographical reasons.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68649 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2026-01-23 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of EBV DNA testing, P85-Ab testing and the two-antibody method testing | At screening, 3 years and 10 years thereafter.
  To investigate whether plasma EBV DNA testing or the P85-Ab testing can achieve higher sensitivity than the current standard two-antibody method testing while maintaining specificity in NPC screening. Sensitivity refers to the proportion of actual positive cases (true positives) correctly identified by a test.
Sensitivity and positive predictive value (PPV) of the two-step method, single-step method and each single screening testing. | At screening, 3 years and 10 years thereafter.
  To determine whether two-step method can further improve the positive predictive value (PPV) while maintaining non-inferior sensitivity. PPV refers to the proportion of positive test results that are true positives. Sensitivity refers to the proportion of actual positive cases (true positives) correctly identified by a test.

SECONDARY OUTCOMES:
Negative predictive value (NPV) | At screening, 3 years and 10 years thereafter.
  NPV refers to the proportion of positive negative results that are true negatives.
Early diagnosis rate of nasopharyngeal carcinoma | At screening, 3 years and 10 years thereafter.
  The proportion of nasopharyngeal carcinoma patients diagnosed at stages I and II according to the 9th version of AJCC TNM system.
Number needed to screen (NNS) | At screening, 3 years and 10 years thereafter.
  NNS refers to the amount of screening participants to identify one nasopharyngeal carcinoma case.
Nasopharyngeal Carcinoma Death Rates | At screening, 3 years and 10 years thereafter.
  Nasopharyngeal Carcinoma deaths confirmed in participants by a death review committee if available, otherwise by death certificate. Rate is the number of deaths divided by person years of follow-up in the study.
Death Rates From All Causes | At screening, 3 years and 10 years thereafter.
  Deaths confirmed in participants by a death review committee if available, otherwise by death certificate. Rate is the number of deaths divided by person years of follow-up in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-yuan Chen, MD, PhD, Study Chair — Sun Yat-sen University
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China